CLINICAL TRIAL: NCT04494217
Title: The Influence of Phototherapy Lights on the Measurement of Oxygen Saturation With Pulse Oximeter in Newborns.
Brief Title: The Effect of Phototherapy Treatment on Oxygen Saturation Measurement in Newborns
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, H. Tolga Çelik, MD, Assistant Professor in Neonatology, Hacettepe University
Other Study IDs: 18815
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hyperbilirubinemia, Neonatal Indirect
Keywords: pulse oximeter, phototherapy, newborn
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This will be a prospective clinical study conducted with the approval of the Clinical Research Ethics Committee.

The influence of phototherapy lights on the accuracy of pulse oximetry will be investigated.

DETAILED DESCRIPTION:
Each patient's oxygen saturation will be measured non-invasively via a nondisposable polyethylene neonatal probe taped to the infant's palm, toe, or dorsum of the foot. The probe will be connected to an Massimo Rad97 pulse oximeter that is standardized at the factory. It runs through an automatic systems check when turned on and needs no further calibration before being used. The oxygen saturation measurements will be considered valid when there will be a normal plethysmographic waveform, a fullscale signal strength bar, and a stable heart rate closely approximating an independent electrocardiographic (ECG) pulse rate. The pulse oximeter works by using the technology of plethsmography which allows the detection of an arterial pulse) with oximetry (which measures oxygen saturation at specific wavelengths). The pulse oximeter will be placed on each infant as already described. After a stable pulse oximeter reading was obtained, the value will be recorded ("before") and then the probe will be covered with a standard disposable diaper, shiny side up. When the reading stabilized, the value will be recorded ("during") and then the diaper will be removed.

ELIGIBILITY:
Inclusion Criteria:

* newborn babies (0-28 days)
* to be treated in the Hacettepe University Children's Hospital Neonatal Intensive Care Unit
* receiving phototherapy treatment

Exclusion Criteria:

* Newborn babies with any diseases that affect oxygen saturation including congenital heart disease, chromosomal disease, inborn error of metabolism, anemia, circulatory disorder, hypovolemia or hydrops fetalis

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborn babies who are receiving phototherapy for indirect hyperbilirubinemia in the NICU of the Hacettepe University will be included in the study following the obtaining of informed consent by their parents/guardian.
  The oxygen saturation of all babies receiving inpatient treatment in the NICU is routinely monitored with a pulse oximeter. In this study, the oxygen saturation of the newborns receiving phototherapy will be recorded.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Percent Oxygen Saturation Before and During Covering Oximeter Probe | The two data (''before'' and ''during'') will be recorded consecutively for each infant, when the reading stabilize. All measurements will be completed wiithin 6 months according to the study protocol calendar.
  The two data points (percent oxygen saturation before and during covering of oximeter probe) for each patient will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vreman HJ, Wong RJ, Stevenson DK. Phototherapy: current methods and future directions. Semin Perinatol. 2004 Oct;28(5):326-33. doi: 10.1053/j.semperi.2004.09.003. PMID 15686263
- [Background] Zubrow AB, Henderson GW, Imaizumi SO, Pleasure JR. Pulse oximetry in sick premature infants and the effects of phototherapy and radiant warmers on the oxygen saturation readout. Am J Perinatol. 1990 Jan;7(1):75-8. doi: 10.1055/s-2007-999451. PMID 2294914